CLINICAL TRIAL: NCT04248933
Title: Peer-Delivered Behavioral Activation Intervention to Improve Adherence to MAT Among Low-Income, Minority Individuals With OUD - Pilot Phase
Brief Title: Peer-Delivered Behavioral Activation for Methadone Adherence - Pilot Phase
Acronym: HEAL Together
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: University of Maryland, Baltimore (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jessica Magidson, Associate Professor, University of Maryland, College Park
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1531148; R61AT010799 (NIH)
Record Dates: First submitted 2020-01-15; First posted 2020-01-30 (Actual); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Substance Use; Substance Use Disorders; Opioid-use Disorder; Peer Delivered; Medication for Opioid Use Disorder (MOUD); Methadone Treatment; Retention in Care; Behavioral Activation
Keywords: Substance-Related Disorders; Medication Treatment for Opioid Use Disorder; Opioid Crisis; Epidemic, Opioid; Opioid Addiction; Treatment Adherence; Retention in Care
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer-Delivered Behavioral Activation ("Peer Activate") (Experimental): Participants received a peer recovery specialist-delivered behavioral activation (BA) intervention ("Peer Activate") to address barriers to retention in methadone treatment and increase substance-free, positive reinforcement to support retention.
  Interventions: Behavioral: Peer-Delivered Behavioral Activation (Peer Activate)

INTERVENTIONS:
Behavioral: Peer-Delivered Behavioral Activation (Peer Activate) — The Peer Activate intervention consisted of weekly one-hour BA sessions led by a peer recovery specialist (PRS) for up to 12 weekly sessions, with the first five being the core treatment sessions and content, and the subsequent seven designed to reinforce core content. In these sessions, participants received individualized support in learning skills to assist in their retention and persistence in methadone treatment and were guided through exercises aimed at incorporating substance-free, rewarding activities into their daily life.

SUMMARY:
The purpose of this study is to evaluate the feasibility and effectiveness of a peer-led, brief, behavioral intervention to improve adherence to medication for opioid use disorder (MOUD) among low-income, minoritized individuals living with opioid use disorder (OUD) in Baltimore, Maryland. The intervention is based on behavioral activation (BA) and is specifically designed to be implemented by a trained peer recovery specialist. In this pilot trial, the investigators will evaluate the feasibility, acceptability, and fidelity of this approach (implementation outcomes) and preliminary effectiveness on methadone treatment retention at three months.

DETAILED DESCRIPTION:
Opioid use disorder (OUD) disproportionately affects low-income, racial/ethnic minorities (Stahler, 2018). MOUD is efficacious for treating OUD. However, adherence to MOUD is often low, which includes poor treatment retention, especially among low-income, racial/ethnic minority individuals (Stahler, 2018;Williams, 2017). This may be due to barriers such as stigma, challenges navigating services, housing instability, fluctuating motivation and readiness, and other structural and psychosocial factors (Timko, 2016;Carroll, 2015).

Peer recovery specialists (PRSs) may be uniquely suited to address these barriers to retention (Jack, 2017;Bassuk, 2016). PRSs are trained individuals who have a personal, lived experience with substance use. Using their lived experience, PRSs can support individuals with OUD to stay retained in care. Rapid increases in the use of PRSs nationwide demonstrate the appeal of employing PRSs as a potentially sustainable solution to support the behavioral treatment needs in OUD care. Yet, few evidence-based interventions have been evaluated for PRS delivery to promote MOUD retention.

Prior research has been inconclusive regarding psychosocial interventions to support MOUD retention (Timko, 2016; Carroll, 2017). Reinforcement-based approaches, such as contingency management, have empirical support for improving MOUD retention, but also can have low adoption in community settings due to organizational and provider barriers, including cost in medically underserved areas (Timko, 2016; Carroll, 2017; Carroll, 2015). Successful interventions need to be not only effective in improving MOUD retention, but also be feasible and sustainable to deliver for underserved populations.

Behavioral activation (BA) may be a feasible, scalable, reinforcement-based approach for improving MOUD retention for low-income, minority individuals with OUD (Magidson, 2011). Originally developed as an efficacious treatment for depression, BA aims to increase positive reinforcement by promoting engagement in adaptive, valued behaviors (Lejuez, 2011). By targeting increases in positive reinforcement, BA has been effective in improving substance use disorder (SUD) treatment retention and preventing future relapse among low-income, minority individuals with SUD. Further, BA has improved medication adherence (i.e., for HIV) among low-income, minority populations with SUD, as well as depression, which may also be a barrier to MOUD retention. Importantly for implementation, BA has previously been implemented in low-resource settings (largely internationally) using lay health workers (e.g., peers, community health workers). However, to date, prior work has yet to evaluate a PRS-delivered BA intervention to support MOUD retention.

This study builds upon formative work to adapt and evaluate PRS-delivered BA to support MOUD retention for low-income, minoritized individuals initiating methadone at an outpatient, opioid treatment program in a medically underserved community in Baltimore, Maryland (Magidson, 2011; Magidson, 2018; Satinsky, 2020). The current study has three phases, the first being formative, qualitative work, to adapt the proposed treatment approach. The second phase is a pilot trial (current phase). The pilot trial is an open-label, Type 1 hybrid effectiveness-implementation trial assessing the feasibility, acceptability, and fidelity (implementation outcomes) of a PRS-delivered BA intervention for MOUD retention in methadone treatment, and evaluating retention in the methadone program at three months (primary effectiveness outcome).

ELIGIBILITY:
Inclusion Criteria:

* Initiated methadone at the study site or demonstrated challenges with methadone adherence in the past three months (e.g., at least one indicator of a missed methadone dose)
* Minimum of 18 years old

Exclusion Criteria:

* Demonstrating active, unstable or untreated psychiatric symptoms, including mania and/or psychosis that would interfere with study participation
* Inability to understand the study and provide informed consent in English
* Positive pregnancy status at enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica F Magidson, PhD, Principal Investigator — Assistant Professor
Locations (2):
- United States (2):
  - University of Maryland Baltimore Drug Treatment Center, Baltimore, Maryland
  - University of Maryland, College Park, College Park, Maryland

IPD SHARING:
Plan to Share IPD: Yes
After all primary analyses are complete, de-identified data will be available per request of outside individual.

REFERENCES:
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Stahler GJ, Mennis J. Treatment outcome disparities for opioid users: Are there racial and ethnic differences in treatment completion across large US metropolitan areas? Drug Alcohol Depend. 2018 Sep 1;190:170-178. doi: 10.1016/j.drugalcdep.2018.06.006. Epub 2018 Jul 11. PMID 30041092
- [Background] Williams AR, Nunes E, Olfson M. To battle the opioid overdose epidemic, deploy the 'Cascade of Care' model. Health Affairs Blog 2017 doi: 10.1377/hblog20170313.059163. Epub: 2017 Mar 13.
- [Background] Timko C, Schultz NR, Cucciare MA, Vittorio L, Garrison-Diehn C. Retention in medication-assisted treatment for opiate dependence: A systematic review. J Addict Dis. 2016;35(1):22-35. doi: 10.1080/10550887.2016.1100960. Epub 2015 Oct 14. PMID 26467975
- [Background] Jack HE, Oller D, Kelly J, Magidson JF, Wakeman SE. Addressing substance use disorder in primary care: The role, integration, and impact of recovery coaches. Subst Abus. 2018;39(3):307-314. doi: 10.1080/08897077.2017.1389802. Epub 2017 Nov 13. PMID 28991516
- [Background] Bassuk EL, Hanson J, Greene RN, Richard M, Laudet A. Peer-Delivered Recovery Support Services for Addictions in the United States: A Systematic Review. J Subst Abuse Treat. 2016 Apr;63:1-9. doi: 10.1016/j.jsat.2016.01.003. Epub 2016 Jan 13. PMID 26882891
- [Background] Carroll KM, Weiss RD. The Role of Behavioral Interventions in Buprenorphine Maintenance Treatment: A Review. Am J Psychiatry. 2017 Aug 1;174(8):738-747. doi: 10.1176/appi.ajp.2016.16070792. Epub 2016 Dec 16. PMID 27978771
- [Background] Carroll KM. Lost in translation? Moving contingency management and cognitive behavioral therapy into clinical practice. Ann N Y Acad Sci. 2014 Oct;1327(1):94-111. doi: 10.1111/nyas.12501. Epub 2014 Sep 9. PMID 25204847
- [Background] Magidson JF, Gorka SM, MacPherson L, Hopko DR, Blanco C, Lejuez CW, Daughters SB. Examining the effect of the Life Enhancement Treatment for Substance Use (LETS ACT) on residential substance abuse treatment retention. Addict Behav. 2011 Jun;36(6):615-623. doi: 10.1016/j.addbeh.2011.01.016. Epub 2011 Jan 21. PMID 21310539
- [Background] Magidson JF, Regan S, Jack HE, Wakeman SE. Reduced hospitalizations and increased abstinence six months after recovery coach contact. American Society of Addiction Medicine. San Diego, CA, 2018.
- [Background] Satinsky EN, Doran K, Felton JW, Kleinman M, Dean D, Magidson JF. Adapting a peer recovery coach-delivered behavioral activation intervention for problematic substance use in a medically underserved community in Baltimore City. PLoS One. 2020 Jan 31;15(1):e0228084. doi: 10.1371/journal.pone.0228084. eCollection 2020. PMID 32004328
- [Background] Lejuez CW, Hopko DR, Acierno R, Daughters SB, Pagoto SL. Ten year revision of the brief behavioral activation treatment for depression: revised treatment manual. Behav Modif. 2011 Mar;35(2):111-61. doi: 10.1177/0145445510390929. PMID 21324944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at a community-based opioid treatment program (OTP) in Baltimore City between October 2020 and August 2021. The OTP program is certified by the Maryland Department of Health Commission on Accreditation of Rehabilitation Facilities and currently serves approximately six hundred active patients receiving methadone treatment. Participants were recruited through word-of-mouth, flyers left at methadone dosing, on-site recruitment tables (outdoor and indoor), and staff referral.
Groups:
- Peer-Delivered Behavioral Activation ("Peer Activate"): Participants received a peer recovery specialist-delivered behavioral activation (BA) intervention ("Peer Activate") to address barriers to retention in methadone treatment and increase substance-free, positive reinforcement to support retention.
  The Peer Activate intervention consisted of weekly one-hour BA sessions led by a peer recovery specialist (PRS) for up to 12 weekly sessions, with the first five being the core treatment sessions and content, and the subsequent seven designed to reinforce core content. In these sessions, participants received individualized support in learning skills to assist in their retention and persistence in methadone treatment and were guided through exercises aimed at incorporating substance-free, rewarding activities into their daily life.
Period: Overall Study
Arm/Group | Peer-Delivered Behavioral Activation ("Peer Activate")
Started | 37 (N = 37 participants were consented and determined to be eligible upon the completion of the baseline assessment.)
Initiated Peer Activate | 32 (Thirty-seven individuals were enrolled in the open-label trial (intent-to-treat sample), with the goal of reaching a minimum of n = 30 Peer Activate initiators (i.e., defined as completing ≥ 1 Peer Activate session). Of the N = 37 intent-to-treat sample, 32 participants completed at least one Peer Activate session and were defined as the "treatment initiator "group.)
Completed Peer Activate Completers (>= 4 Sessions) | 26 (Thirty-two individuals initiated the Peer Activate intervention, with the goal of reaching a minimum of n = 24 completers (i.e., defined as completing ≥ four Peer Activate sessions). Of the N = 32 "treatment initiators" group, 26 participants completed at least four Peer Activate sessions and were defined as the "treatment completer" group.)
Completed | 26 (Twenty-six participants completed the post-treatment assessment. This includes n=3 who completed the post-treatment assessment prior to the 4th session and excludes n=3 who completed 4 Peer Activate sessions but did not complete a post-treatment assessment.)
Not Completed | 11
Not completed — Lost to Follow-up | 9
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Peer-Delivered Behavioral Activation ("Peer Activate")
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.81 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 11
  More than one race | 6
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: MOUD Retention Rate: % of Patients Retained at 3 Months
Description: Percent of patients retained in MOUD treatment at three months (i.e. still engaged in care) after intervention enrollment.
Time Frame: Measured daily from intake to post-treatment (approximately 12-weeks)
Population: Verification of methadone retention at the study site and/or outside methadone treatment programs was able to be established for 94.6% of participants (35/37) at monthly intervals (one, two, and three months post-intervention). Two participants were coded as missing, as we were unable to verify their status at an outside treatment program after being transferred.
Measure: Count of Participants; unit: Participants
Arm/Group | Peer-Delivered Behavioral Activation ("Peer Activate")
Number analyzed (Participants) | 35
Participants | 31

2. Primary Outcome: Intervention Feasibility: % of Patients Who Agree to Participate in the Intervention
Description: Feasibility, defined as the suitability and practicability of the approach, was measured quantitatively as the % of patients who agreed to participate in the intervention.
Time Frame: Assessed between the baseline assessment and the acute outcome (approximately 12-weeks post-baseline assessment/ post-treatment assessment)
Population: Enrolled in the open-label trial (intent-to-treat sample)
Measure: Count of Participants; unit: Participants
Arm/Group | Peer-Delivered Behavioral Activation ("Peer Activate")
Number analyzed (Participants) | 37
Participants | 32

3. Secondary Outcome: Intervention Acceptability: % of Patients Who Attend ≥75% Sessions
Description: Acceptability, defined as satisfaction with or tolerability of the proposed approach, was measured quantitatively by session attendance. Specifically, we measured the % of patients who attended ≥75% of core intervention sessions.
Time Frame: as for outcome 2
Population: Participants who initiated the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Peer-Delivered Behavioral Activation ("Peer Activate")
Number analyzed (Participants) | 32
Participants | 26

4. Secondary Outcome: Intervention Fidelity: Percentage of Intervention Components Delivered by Peer as Intended
Description: Fidelity, defined as the delivery of the intervention as intended, was measured based on PRS adherence to the intervention delivery. A random selection of 20% of sessions was rated for fidelity, and we assessed the % of intervention components delivered as intended.
Time Frame: as for outcome 2
Population: We selected a random 20% of recorded intervention sessions across individuals who initiated the intervention (n=32), with some additional sessions re-assigned when the originally selected sessions were not completed and additional sessions coded early on in the trial for training purposes.
Measure: Mean (Standard Deviation); unit: Percentage fidelity to treatment
Units Other Than Participants: intervention session recordings
Arm/Group | Peer-Delivered Behavioral Activation ("Peer Activate")
Number analyzed (Participants) | 32
Number analyzed (intervention session recordings) | 81
Percentage fidelity to treatment | 87.9 (18.0)

5. Other Pre Specified Outcome: Change in Opioid Use
Description: Assessed point prevalence of indicators of opioid use in urinalysis.
Time Frame: as for outcome 2
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Methadone Use
Description: Assessed point prevalence of indicators of methadone use in urinalysis.
Time Frame: as for outcome 2
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Depressive Symptoms
Description: Patient Health Questionnaire-8 (PHQ-8). Possible score of 0 - 24, with higher scores indicating more depressive symptoms.
Time Frame: as for outcome 2
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed between the baseline assessment and the acute outcome (approximately 12 weeks post-baseline assessment/ post-treatment assessment).
Arm/Group | Peer-Delivered Behavioral Activation ("Peer Activate")
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 11/37
Other Adverse Events (participants affected / at risk) | 5/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peer-Delivered Behavioral Activation ("Peer Activate") (N=37)
Hospitalization (Injury, poisoning and procedural complications) | 5 (5)
Hospitalization (Infections and infestations) | 2 (2)
Hospitalization (Psychiatric disorders) | 1 (1)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalization (General disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peer-Delivered Behavioral Activation ("Peer Activate") (N=37)
Medical event (Injury, poisoning and procedural complications) | 2 (2)
Medical event (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Medical event (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT04248933/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT04248933/SAP_001.pdf